CLINICAL TRIAL: NCT05125965
Title: Contribution of Cardiac MRI in the Early Diagnosis of Myocarditis Induced by Immunotherapy
Acronym: MEDIIMYO
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Centre Chirurgical Marie Lannelongue (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: ID RCB : 2021-A01656-35
Record Dates: First submitted 2021-11-02; First posted 2021-11-18 (Actual); Last update posted 2021-11-18 (Actual); Status verified 2021-11

CONDITIONS: Myocarditis
Keywords: anti-cancer immunotherapy; cardiac autoimmune diseases; Myocarditis
MeSH Terms: conditions — Myocarditis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patient undergoing immunotherapy with an indication for cardiac MRI (Experimental): Patient undergoing immunotherapy with an indication for cardiac MRI for suspected myocarditis or myocarditis or other cardiovascular complications
  Interventions: Other: additional time for the MRI

INTERVENTIONS:
Other: additional time for the MRI — 3 additional minutes to perform the MRI

SUMMARY:
Anti-cancer immunotherapy, one of the therapeutic revolutions of recent years. It is based on the use of antibodies that block immune system checkpoints that have been hijacked by cancer cells to benefit themselves. Blocking these checkpoints, such as PD-1, unleashes the action of anti-cancer T cells that can then destroy the tumor. The efficacy of these targeted therapies is significant, with an average 40% response rate in patients with metastatic cancers.Immune checkpoint inhibitors (ICIs) are becoming a 1st line therapy in many oncology indications due to their therapeutic line in many oncology indications due to their favorable effect on the prognosis of various prognosis of various cancers Since checkpoints play a key role in controlling the intensity and duration of an immune response, their immune response, therefore, their inhibition exposes to adverse inflammatory or autoimmune effects inflammatory or autoimmune adverse effects that can be severe and sometimes lethal.Most side effects of ICIs occur within the first few months after initiation of treatment. The toxicity of immunotherapy is immunological, all organs including the heart can be including the heart, can be affected.

Cardiac autoimmune involvement in ICIs can involve the myocardium, pericardium, and/or vascular endothelium. These entities may be interrelated or, on the contrary, isolated.

In the last 5 years, the number of described cases of myocarditis associated with ICIstreatment has increased. Their incidence remains low, estimated between 0.5 and 2%. This probably represents the most serious cardiovascular complication, as the mortality attributed to it reaches almost 50%.

In recent years MRI has become very important in the noninvasive diagnosis of acute myocarditis. The latest update of the Lake Louise criteria in 2018 has thus confirmed cardiac MRI in its first place among noninvasive examinations for the diagnosis of myocarditis with a sensitivity of 87.5%, a specificity of 96.2%, and a positive predictive value of 97.2%.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing immunotherapy with an indication for cardiac MRI for suspected myocarditis or other cardiovascular complications
* Patient over 18 years of age
* Patient affiliated to a health insurance plan
* Patient who has given free, informed and oral consent

Exclusion Criteria:

* Contraindication to immunotherapy
* Pregnant or breastfeeding patient (if applicable)
* Contraindication to cardiac MRI

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2021-11-15 (Estimated); Primary Completion 2023-11-15 (Estimated); Study Completion 2024-11-15 (Estimated)

PRIMARY OUTCOMES:
cardiac MRI | 1 day
  ejection fraction

CONTACTS AND LOCATIONS:
Locations (1):
- Centre Chirurgical Marie Lannelongue, Le Plessis-Robinson, France